CLINICAL TRIAL: NCT07110402
Title: Clinical and Comparative Evaluation of Treatment Results for Osteoarthritis of the Knee in the Form of Chondromalacia of the Articular Cartilage Treated in the Arthroscopic Technique With the Use of: Autogenous Transplant of Fragmented Adipose Tissue Taken From Abdominal Integuments, PRP GF (Platelet-rich Plasma With Growth Factors), Mesenchymal Cells Centrifuged From Bone Marrow Cells Taken From the Iliac Crest, Hyaluronic Acid - Low Molecular Weight, Hyaluronic Acid - Cross-linked
Brief Title: Evaluation of Treatment of Osteoarthritis of the Knee in the Form of Chondromalacia of the Articular Cartilage Treated in the Arthroscopic Technique With the Use of:Autogenous Transplantation of Fragmented Adipose Tissue,PRP GF,Mesenchymal Cells,Hyaluronic Acid-low Molecular Weight and Cross-linked
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: eMKa MED Medical Center (Other)
Collaborators: Wroclaw Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KB-633/2022
Record Dates: First submitted 2025-07-23; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Osteoarthritis, Knee; Chondral Defect; Chondromalacia, Left Knee; Chondromalacia, Right Knee; Articular Cartilage Disorder of Knee
Keywords: Cartilage; Damage; Chondral defect; Chondromalacja; Techniques; Articular Cartilage Treated; Autogenous Transplant; PRP GF; Hyaluronic Acid; Mesenchymal Cells
MeSH Terms: conditions — Osteoarthritis, Knee; Cartilage Diseases | interventions — Intercellular Signaling Peptides and Proteins

STUDY DESIGN:
Intervention Model Description: 1. Autogenous transplant of fragmented adipose tissue taken from abdominal integuments - (MyStem, Lipogems, Arthrex)
  2. PRP GF (platelet-rich plasma with growth factors) (Ycellbio, ACP Arthrex, Neoregen, FrankPharma)
  3. Mesenchymal cells centrifuged from bone marrow cells taken from the iliac crest - (Harvest, Arthrex)
  4. Hyaluronic acid - low molecular weight (Synvisc, Biolevox, ArtiAidPlus)
  5. Hyaluronic acid - cross-linked Arti Aid Plus, Synovial, Durolain, StavOn, Collagenu - Guna, Orthokine.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Autogenous transplant of fragmented adipose tissue taken from abdominal integuments (Experimental): Treatment of chondromalacia of the cartilage in the knee joint with the use of autogenous graft of fragmented adipose tissue taken from the abdominal wall - MyStem, Lipogems, Arthrex.
  Interventions: Procedure: Autogenous transplant of fragmented adipose tissue taken from abdominal integuments
- PRP GF (platelet-rich plasma with growth factors) (Experimental): Treatment of chondromalacia of the cartilage in the knee joint with the use of PRP GF (platelet-rich plasma with growth factors: Ycellbio, ACP Arthrex, Neoregen, PhankPharma).
  Interventions: Procedure: PRP GF (platelet-rich plasma with growth factors)
- Mesenchymal cells centrifuged from bone marrow cells taken from the iliac crest (Experimental): Treatment of cartilage chondromalacia in the knee joint using mesenchymal cells centrifuged from bone marrow cells taken from the iliac crest - (Harvest, Arthrex),
  Interventions: Procedure: Mesenchymal cells centrifuged from bone marrow cells taken from the iliac crest
- Hyaluronic acid - low molecular weight (Experimental): Treatment of chondromalacia of the cartilage in the knee joint with the use of Hyaluronic Acid - low molecular weight (Synvisc, Biolevox, ArtiAidPlus).
  Interventions: Procedure: Hyaluronic acid - low molecular weight
- Hyaluronic acid - cross-linked (Experimental): Treatment of chondromalacia of the cartilage in the knee joint with the use of cross-linked Hyaluronic Acid Arti Aid Plus, Synovial, Durolain, StavOn, Collagenu - Guna, Orthokine.
  Interventions: Procedure: Hyaluronic acid - cross-linked

INTERVENTIONS:
Procedure: Autogenous transplant of fragmented adipose tissue taken from abdominal integuments — Treatment of chondromalacia of the cartilage in the knee joint by arthroscopic technique with the use of autogenous graft of fragmented adipose tissue taken from the abdominal wall.
  Arms: Autogenous transplant of fragmented adipose tissue taken from abdominal integuments
Procedure: PRP GF (platelet-rich plasma with growth factors) — Treatment of chondromalacia of the cartilage in the knee joint by arthroscopic technique with the use of PRP GF (platelet-rich plasma with growth factors)
  Arms: PRP GF (platelet-rich plasma with growth factors)
Procedure: Mesenchymal cells centrifuged from bone marrow cells taken from the iliac crest — Treatment of cartilage chondromalacia in the knee joint by arthroscopic technique using mesenchymal cells centrifuged from bone marrow cells taken from the iliac crest
  Arms: Mesenchymal cells centrifuged from bone marrow cells taken from the iliac crest
Procedure: Hyaluronic acid - low molecular weight — Treatment of chondromalacia of the cartilage in the knee joint with the use of Hyaluronic Acid - low molecular weight
  Arms: Hyaluronic acid - low molecular weight
Procedure: Hyaluronic acid - cross-linked — Treatment of chondromalacia of the cartilage in the knee joint by arthroscopic technique with the use of cross-linked Hyaluronic Acid Arti Aid Plus, Synovial, Durolain, StavOn, Collagenu
  Arms: Hyaluronic acid - cross-linked

SUMMARY:
The main objective of the research project is to evaluate the results of the treatment of chondromalacia of the cartilage in the knee joint with the use of: autogenous transplantation of fragmented adipose tissue taken from the abdominal wall - (MyStem, Lipogems, Arthrex).

PRP GF (platelet-rich plasma with growth factors) (Ycellbio, ACP Arthrex, Neoregen, FrankPharma), Mesenchymal cells centrifuged from bone marrow cells taken from the iliac crest - (Harvest, Arthrex), Hyaluronic acid - low molecular weight (Synvisc, Biolevox, ArtiAidPlus), Hyaluronic acid - cross-linked Arti Aid Plus, Synovial, Durolain, StavOn, Collagen - Guna, Orthokine.

The specific objectives are: to compare the results of treatment of analogous zones of cartilage defects in the knee joint obtained in the study groups using two methods: microfractures and microfractures with simultaneous intra-articular injection of autogenous cartilage graft and PRP GF (Auto Cart-Arthrex method). The results for the operated limb in both groups will be compared both between the groups and with the results of clinical and biomechanical tests for the non-operated limbs.

DETAILED DESCRIPTION:
The study will be prospective, randomized. The study groups will consist of 30 people with damage to analogous cartilage zones of the knee joint qualified for arthroscopic treatment.

After surgery, patients will be improved according to the same rehabilitation protocol.

The follow-up examination will include: subjective assessment and clinical examination on day 1, then after 3 and 6 months, MRI imaging, ultrasound after 6 months, biomechanical examination after 3 and 6 months.

A detailed interview will be conducted in the study groups, supplemented with pain assessment on the 1st day after the procedure using the Visual Analogue Scale (VAS), Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), then with the TAS activity level scale (TAS). Tegner Activity Level Scale), three parts of the 2000 International Knee Documentation Committee (2000 IKDC) questionnaire: Demographic Form, Current Health Assessment Form, percentage of drugs used acute treatment initiation, withdrawal rates due to knee pain, knee range of motion, and adverse events.

The MRI examination will be carried out on a 1.5 Tesla apparatus, the ultrasound examination on a apparatus with the option of elastometry and BMI.

Measurements of the range of motion of the knee joint, measurements of the circumference of the knee joint and thigh, measurements of the torques of the extensor and flexor muscles of the knee joint as well as the muscles responsible for the internal and external rotation of the lower leg relative to the thigh in the knee joint in static and isokinetic conditions, measurements of proprioception on the Biodex 4 measuring stand System, measurements of gait kinetics and kinematics using the BTS Smart optoelectronic system for three-dimensional movement analysis and two Kistler strain gauge platforms, as well as the squat test.

ELIGIBILITY:
Inclusion Criteria:

* Surgery for ACL damage to the knee joint;
* Arthroscopic surgery;
* No prior knee surgical interventions;
* No additional pathologies in this anatomical area;
* Informed consent of the patient to participate in the study.

Exclusion Criteria:

* Previous surgical interventions in the examined anatomical area;
* Additional pathologies in this area identified as part of preoperative diagnostics;
* Damage to the second knee joint;
* Failure to comply with the rigor of the same rehabilitation treatment protocol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2022-12-12 (Actual); Primary Completion 2024-12-12 (Actual); Study Completion 2024-12-12 (Actual)

PRIMARY OUTCOMES:
Tegner Activity Level Scale (TAS) | 1 day
  The Tegner Activity Scale (TAS) aims to provide a standardized method in determining the level of activity prior to injury and level of activity post injury that can be documented on a numerical scale.
  The Tegner activity scale is a one-item score that graded activity based on work and sports activities on a scale of 0 to 10. Zero represents disability because of knee problems and 10 represents national or international level soccer.
Tegner Activity Level Scale (TAS) | 3 months after procedure
  The Tegner Activity Scale (TAS) aims to provide a standardized method in determining the level of activity prior to injury and level of activity post injury that can be documented on a numerical scale.
  The Tegner activity scale is a one-item score that graded activity based on work and sports activities on a scale of 0 to 10. Zero represents disability because of knee problems and 10 represents national or international level soccer.
Tegner Activity Level Scale (TAS) | 6 months after procedure
  The Tegner Activity Scale (TAS) aims to provide a standardized method in determining the level of activity prior to injury and level of activity post injury that can be documented on a numerical scale.
  The Tegner activity scale is a one-item score that graded activity based on work and sports activities on a scale of 0 to 10. Zero represents disability because of knee problems and 10 represents national or international level soccer.
Visual Analogue Score (VAS) | 1 day
  In this method, the examined person marks a point on a line with a length of (for example) 10 cm, where the value 0 is assigned to the complete absence of pain, and the value 10 to the strongest pain imaginable.
Visual Analogue Score (VAS) | 3 months after procedure
  In this method, the examined person marks a point on a line with a length of (for example) 10 cm, where the value 0 is assigned to the complete absence of pain, and the value 10 to the strongest pain imaginable.
Visual Analogue Score (VAS) | 6 months after procedure
  In this method, the examined person marks a point on a line with a length of (for example) 10 cm, where the value 0 is assigned to the complete absence of pain, and the value 10 to the strongest pain imaginable.
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | 1 day
  The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) is defined as a disease-specific instrument used for assessing quality of life, particularly focusing on activity limitation in individuals with osteoarthritis.
  The WOMAC consists of three subscales and has a total possible score range of 0 to 96: pain (five questions), stiffness (two questions), and physical function (17 questions). The subscale scores can vary, with pain ranging from 0 to 20 points; stiffness, 0 to 8 points; and physical function, 0 to 68 points.
  Lower scores indicate better health status (less pain, stiffness, and functional limitations), while higher scores represent worse outcomes ( worse pain, stiffness, and functional limitations).
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | 3 months after procedure
  The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) is defined as a disease-specific instrument used for assessing quality of life, particularly focusing on activity limitation in individuals with osteoarthritis. The WOMAC consists of three subscales and has a total possible score range of 0 to 96: pain (five questions), stiffness (two questions), and physical function (17 questions). The subscale scores can vary, with pain ranging from 0 to 20 points; stiffness, 0 to 8 points; and physical function, 0 to 68 points. Lower scores indicate better health status (less pain, stiffness, and functional limitations), while higher scores represent worse outcomes ( worse pain, stiffness, and functional limitations).
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | 6 months after procedure
  The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) is defined as a disease-specific instrument used for assessing quality of life, particularly focusing on activity limitation in individuals with osteoarthritis. The WOMAC consists of three subscales and has a total possible score range of 0 to 96: pain (five questions), stiffness (two questions), and physical function (17 questions). The subscale scores can vary, with pain ranging from 0 to 20 points; stiffness, 0 to 8 points; and physical function, 0 to 68 points. Lower scores indicate better health status (less pain, stiffness, and functional limitations), while higher scores represent worse outcomes ( worse pain, stiffness, and functional limitations).
IKDC SUBJECTIVE KNEE EVALUATION FORM | 1 day
  Interpreted as a measure of function, such that higher scores represent higher levels of function and lower levels of symptoms. A score of 100 is interpreted to mean no limitation with sporting activities or daily living and the complete absence of symptoms.
IKDC SUBJECTIVE KNEE EVALUATION FORM | 3 months after procedure
  Interpreted as a measure of function, such that higher scores represent higher levels of function and lower levels of symptoms. A score of 100 is interpreted to mean no limitation with sporting activities or daily living and the complete absence of symptoms.
IKDC SUBJECTIVE KNEE EVALUATION FORM | 6 months after procedure
  Interpreted as a measure of function, such that higher scores represent higher levels of function and lower levels of symptoms. A score of 100 is interpreted to mean no limitation with sporting activities or daily living and the complete absence of symptoms.
Biomechanical examination | 3 months after procedure
  On the Biodex 3 System measuring device
Biomechanical examination | 6 months after procedure
  On the Biodex 3 System measuring device
Magnetic resonance imaging (MRI) of the knee joint | 6 months after procedure
  MRI (1.5 Tesli) will be used to assess the cartilage healing process following arthroscopic surgery. Radiological assessment will include cartilage defect fill, tissue integration, surface smoothness, and signal intensity of repair tissue.
  An imaging appearance indicative of effective healing is interpreted as a better outcome.
Ultrasound examination (USG) of the knee joint | 6 months after procedure
  Ultrasound examination on the apparatus with the option of elastometry will be used to assess postoperative tissue regeneration and intra-articular conditions. USG will be performed using a linear transducer with a frequency of 7-10 MHz. The evaluation will include: cartilage surface regularity and thickness, presence or absence of joint effusion, synovial membrane hypertrophy (synovitis), swelling or inflammatory changes in Hoffa's fat pad, signs of active inflammation.
  An imaging appearance indicative of effective healing is interpreted as a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- eMKa MED Medical Center, Wroclaw, Dolnośląsk, Poland